CLINICAL TRIAL: NCT01974466
Title: Fluid Resuscitation Goal in Early Stage of Severe Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Erzhen Chen, Professor, Ruijin Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RJpancreatitis01; RJpancreatitis01 (Registry Identifier: RuijinH)
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatitis
Keywords: pancreatitis; resuscitation goal
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goal A (Active Comparator): controled fluid therapy: 5~10ml/kg/hr fulfillment of two or more of four criteria:
  1. heart rate <120 beats/min,
  2. mean arterial blood pressure 65-85 mm Hg,
  3. urine output ≥1 ml/kg /h
  4. Hematocrit ≤35%.
  Interventions: Other: Goal A
- Goal B (Other): controled fluid therapy: 5~10ml/kg/hr fulfillment of all of the following criteria:
  1 central venous pressure8-12 mmHg , 2.mean arterial pressure 65-85 mm Hg, 3. urine output ≥0.5 ml/kg/h 4. ScvO2 ≤70%
  Interventions: Other: Goal B

INTERVENTIONS:
Other: Goal A — controled fluid therapy：10~5ml/kg/h，crystalloid vs colloid 2:1 resuscitation target： fulfillment of two or more of four criteria:1. HR <120 beats/min, 2.MAP 65-85 mm Hg, 3. urine output ≥1 ml/kg /h 4. HCT ≤35%.
  Other Names: Ruijin pancreatitis goal
  Arms: Goal A
Other: Goal B — controled fluid therapy：10~5ml/kg/h，crystalloid vs colloid 2:1 resuscitation target： fulfillment of all of the following criteria:
  1 CVP 8-12 mmHg , 2.MAP 65-85 mm Hg, 3. urine output ≥0.5 ml/kg/h 4. ScvO2 ≤70%
  Other Names: Sepsis goal
  Arms: Goal B

SUMMARY:
To compare different goals of fluid resuscitation in early stage of acute pancreatitis

DETAILED DESCRIPTION:
With regard to study of sepsis and several studies of SAP demonstrating the deleterious effects of fluid loss and haemoconcentration within the first 24h after admission（or onset of abdominal pain）, early goal-directed fluid resuscitation has the potential of improving outcome also in SAP. But the goal of fluid resuscitation remained controversial.Several criteria of fluid resuscitation had been described. Ours had been described in previous study, and had shown a ideal result with less incidence of abdominal compartment syndrome and higher survival rate. This study aims to determine a better goal of fluid resuscitation in severe acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of pancreatitis: Typical pain increase in serum lipase or amylase 2. Onset of abdominal pain within <=72h before admission 3. moderate severe or severe acute pancreatitis according to Atlanta criteria revisited in 2012 4. Evidence of >= 1 predictor of fluid resuscitation: Haematocrit >44% (male) or >40% (female), respectively Lactate>4mmol/L; heart rate>120bpm; urine <0.5ml/kg/h for 6 hour; Mean arterial pressure>85 or <60 mmHg

Exclusion Criteria:

* 1. Pregnancy 2. New York Heart Association classification >II 3. With pacemaker implantation 4. chronic obstructive pulmonary disease 5. chronic kidney disease 6. Pre-existing disease with life expectancy < 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-09 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28day

SECONDARY OUTCOMES:
intra-abdominal Hypertension | 7 days

OTHER OUTCOMES:
respiratory failure | 14days

CONTACTS AND LOCATIONS:
Overall Officials: Qiang En Mao, PhD, Study Director — Emergency intensive care unit of Ruijin Hospital; Ming zhong, MD, Study Chair — doctor
Locations (1):
- Ruijin, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Mao EQ, Tang YQ, Fei J, Qin S, Wu J, Li L, Min D, Zhang SD. Fluid therapy for severe acute pancreatitis in acute response stage. Chin Med J (Engl). 2009 Jan 20;122(2):169-73. PMID 19187641